CLINICAL TRIAL: NCT03762512
Title: Collection of Donated Placenta for Isolation of Mitochondria for Research and for Future Use in Mitochondrial Augmentation Therapies
Status: Recruiting | Type: Observational
Sponsor: Minovia Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MNV-005
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Placenta will be collected and from these, mitochondrial will be harvested. Mitochondria will be used in mitochondrial augmentation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy pregnant females between the age of 18-45, judged to be medically eligible by the Investigator and the Sponsor's Medical Monitor.
2. Planned elective C-section at weeks 36-41 of pregnancy.
3. Uncomplicated pregnancy as determined by the Investigator.
4. Available Medical History of the donor (diagnosis, diseases, medication etc…)

Exclusion Criteria:

1. Donor is positive for a communicable disease, such as: HBV, HCV, HIV 1&2, WNV, HTLV 1&2, Treponema pallidum, CMV, Chagas, Chlamydia Trachomatis, Neisseria Gonorrhea, or any other tests required by the medical facility, IMoH, FDA, EMA or the Sponsor.
2. Donor is at risk for a communicable disease as assessed by medical history, medical records, physical exam, and the Donor Screening Questionnaire.
3. Donor is at risk for COVID-19 as assessed by medical history, medical records, physical exam, and the COVID-19 Screening Questionnaire.
4. Donor smokes more than one pack of cigarettes a day or drinks more than one alcoholic beverage a day.
5. Donor has taken a medication with potential mitochondrial effects within 2 weeks prior to placental donation, such as valproic acid, aminoglycoside antibiotics, neuromuscular blocking drugs (See Appendix 3).
6. Donor has current or history of malignancy.
7. Donor has current or history of insulin dependent diabetes
8. Donor has current gestational diabetes treated with insulin, or pre-eclampsia.
9. Donor is known to be a carrier of a primary mitochondrial disease.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Must be pregnant
Study Population: Pregnant females giving term birth by C-section
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Placenta donated | immediate
  The purpose of this study is to collect placenta for the production of mitochondria. Therefore, only general measurements are taken such as placenta weight and health of mother during pregnancy. No further intervention or interaction with the mother will occur, and she does not receive any drug product or treatment prior to or after placenta donation.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center Hospital- Tel Hashomer, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No